CLINICAL TRIAL: NCT01038505
Title: Head to Head Comparison of Tacrolimus and Myfortic vs Tacrolimus and Sirolimus Used in Combination in Non-HLA Identical Living Donor Kidney Transplants
Brief Title: Comparison of Tacrolimus and Myfortic Versus Tacrolimus and Sirolimus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lost funding source
Sponsor: University of Miami (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090531
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Living Donor Kidney Transplants Patients
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus and Myfortic (Active Comparator): Immunosuppressive
  Interventions: Drug: Tacrolimus, Myfortic and Sirolimus
- Tacrolimus and Sirolimus (Active Comparator): Immunosuppressive
  Interventions: Drug: Tacrolimus, Myfortic and Sirolimus

INTERVENTIONS:
Drug: Tacrolimus, Myfortic and Sirolimus — Immunosuppressive drugs

SUMMARY:
The investigators center has also analyzed data over the last 7 years from deceased donor (DD) and living donor (LD) kidney transplant recipients who were randomized into 3 immunosuppressive arms between 2000 and 2001. Thus the goal of the investigators study is to reduce the toxic effects of traditional immunosuppressive regimens involving high-dose calcineurin inhibitor agents by comparing low-dose TAC-MYF with low-dose TAC and de novo SRL regimens. In order to minimize exposure to TAC, the investigators center has previously shown favorable outcomes using combination Thymoglobulin and Zenapax (Daclizumab) for anti-lymphocyte induction in the investigator population of patients.

DETAILED DESCRIPTION:
A total of 150 randomized patients divided into 2 arms: 75 patients will be randomized to receive TAC-SRL, and 75 patients to receive TAC-MYF.

ELIGIBILITY:
Inclusion Criteria:

* Non-HLA identical living donor kidney transplant patients

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than a kidney.
* Patient is receiving an ABO incompatible donor kidney.
* Recipient or donor is known seropositive for human immunodeficiency (HIV) or Hepatitis C virus, or Hepatitis B virus antigenemia.
* Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully, or carcinoma in-situ of the cervix that has been treated successfully.
* Patients with significant liver disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range at our center.
* Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with study objectives.
* Patient is currently participating in another clinical trial of an investigational drug in the 30 days prior to transplant.
* Patient will be receiving any immunosuppressive agent other than those prescribed in the study.
* Patient is unable to take medications orally or via nasogastric tube by the morning of the second day following completion of the transplant procedure (i.e., skin closure).
* Patient is receiving or may require Warfarin, Fluvastatin, or herbal supplements during the study.
* Concurrent use of Astemizole, Pimozide, Cisapride, Terfenadine, or Ketoconazole.
* Patient has a known hypersensitivity to Tacrolimus, Thymoglobulin®, IL-2 receptor inhibitor monoclonal antibodies, Rapamune, Myfortic®, or corticosteroids.
* Patient is pregnant or lactating.
* Patients with a screening/baseline (or within 96 hours of transplant) total white blood cell count <4000/mm3; platelet count <100,000/mm3; fasting triglycerides >400 mg/dl (>4.6 mmol/L); fasting total cholesterol >300 mg/dl (>7.8 mmol/L); fasting HDL-cholesterol <30 mg/dl; fasting LDL-cholesterol >200 mg/dl.
* Patient is unlikely to comply with the visits scheduled in the protocol.
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
* If Tacrolimus cannot be instituted for longer than 5 days postoperatively.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the time to initiation of the comparison study | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda Chen, M.D., Principal Investigator — University of Miami